CLINICAL TRIAL: NCT01225991
Title: An Open-label Trial of Milnacipran for the Treatment of Pain in Rheumatoid Arthritis (RA) in Older Adults
Brief Title: Milnacipran for Treatment of Pain in Older Adults With Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Helen Lavretsky, MD, Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAV-MD-10
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Pain, Fatigue, Geriatric, Rheumatoid Arthritis, Milnacipran
MeSH Terms: conditions — Arthritis, Rheumatoid; Pain; Fatigue | interventions — Milnacipran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Milnacipran, active drug, open-label (Experimental): All subjects will be free of antidepressant medications or opiates, or any other medications used to treat pain for at least 2 weeks prior to initiation of dose titration. Patients will be allowed to escalate up to 100 mg a day, or to their maximum tolerated dose in the course of the first week. The stable-dose phase will be a 10-week period during which patients will take medications at the final dose achieved (either 100 mg per day in divided doses, or the maximum tolerated dose of less than 100 mg per day). Final efficacy assessments will be made at the termination visit, and the study medication will be tapered down following 12 weeks of drug treatment.
  Interventions: Drug: Milnacipran

INTERVENTIONS:
Drug: Milnacipran — All subjects will be free of antidepressant medications or opiates, or any other medications used to treat pain for at least 2 weeks prior to initiation of dose titration. Patients will be allowed to escalate up to 100 mg a day: Day 1: 12.5 mg once a day; Days 2-3: 25 mg/day (12.5 mg twice daily); Days 4-7: 50 mg/day (25 mg twice daily); After Day 7: 100 mg/day (50 mg twice daily). The stable-dose phase will be a 10-week period during which patients will take medications at the final dose achieved (either 100 mg per day in divided doses, or the maximum tolerated dose of less than 100 mg per day).
  Other Names: Savella

SUMMARY:
The purpose of this study is to examine the effects of milnacipran for the treatment of pain in rheumatoid arthritis in older adults.

DETAILED DESCRIPTION:
This is a 12-week open-label trial of milnacipran for the treatment of pain in rheumatoid arthritis in older adults. The investigators are interested in the relationship of chronic pain to inflammation, resilience, fatigue, and physical and mental functioning. The investigators anticipate that effective pain reduction will result in improved fatigue, resilience, physical and mental functioning and reduced levels of inflammation. The investigators are seeking to examine this directly in 30 older adults (55 years of age or older) with rheumatoid arthritis who will be using milnacipran for treatment of pain in the absence of clinical major depression. This proposed trial will serve as a pilot study to estimate the effect of the drug on pain and functional outcomes, as well as aid in dose-finding in this population.

ELIGIBILITY:
Inclusion Criteria: Diagnosis. RA subjects will be evaluated by a board certified rheumatologist using revised criteria established by the American College of Rheumatology (ACR). This requires at least four of the following seven criteria: 1) morning joint stiffness; 2) arthritis in 3 or more joint areas; 3) arthritis of hand joints; 4) symmetric arthritis; 5) rheumatoid nodules; 6) presence of serum rheumatoid factor and 7) changes on posteroanterior hand and wrist radiographs. In addition, criteria 1-4 must be present for at least four weeks. Individuals diagnosed with juvenile RA will be excluded.

Inclusion Criteria: Medication Use for RA patients. RA subjects taking disease modifying anti-rheumatic drugs (DMARDs) must be on a stable regime for one month before study and stable throughout study. RA subjects using DMARDs will be categorized as follows: 1) no DMARDs; 2) DMARD monotherapy with sulfasalazine, hydroxychloroquine, minocycline, or azothioprine, 3) DMARD monotherapy with methotrexate or leflunomide, 4) biologic therapy with or without concomitant DMARDs.

Exclusion Criteria: Medical conditions. Subjects will not be eligible for the study based on the following criteria: (1) presence of acute or uncontrolled co-morbid medical conditions not limited to but including cardiovascular (e.g., history of acute coronary event, stroke, uncontrolled HTN) and neurological diseases (e.g., Parkinson's disease), as well as pain disorders; (2) presence of co-morbid inflammatory disorders such as Crohn's disease and ulcerative colitis and other autoimmune disorders; (3) presence of an uncontrolled medical condition that is deemed by the investigators to interfere with the proposed study procedures, or put the study participant at undue risk; (4) presence of chronic infections (e.g. positive purified protein derivative (PPD) test)) due to contraindication of tumor necrosis factor (TNF) antagonist use in these individuals and also because chronic infection can produce elevations in proinflammatory cytokines; (5) presence of an acute infectious illness in the two weeks prior to an experimental session; (6) pregnancy or breast-feeding because of the effects on neuroendocrine systems and sleep; (7) in women, the presence of vasomotor symptoms due to the effects of such symptoms on measures of sleep; (8) use of hormone containing medications including steroids; (9) current and/or regular use of nonsteroidal anti-inflammatory drug (NSAID) medications.

Exclusion Criteria: Psychiatric Disorders. RA subjects with a current or lifetime history of a major Depressive Disorder or other Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) psychiatric disorder (e.g. substance dependence) will be excluded due to the known effects of major depression on pain. Although depressive symptoms can occur in as many as 40% of RA patients, the prevalence of syndromal major depressive disorder is considerably less, and we do not anticipate that exclusion of current or lifetime history of major depressive disorder will substantially alter subject flow. More than 75% of a selected sample of RA subjects at University of California, Los Angeles (UCLA) affiliated clinics does not have a history of co-morbid psychiatric disorder.

Exclusion Criteria: Medication use. Subjects who have used the following medications in the past two months will be excluded from the study: (1) previous use of Nitrogen Mustard, Cyclosporin, Cytotoxin, or Cyclophosphamide; (2) regular use of analgesics such as opioids, (3) regular use of prednisone >10mg of prednisone, (4) psychotropic medications, including selective serotonergic reuptake inhibitors, antidepressants, anxiolytics, hypnotics, sedatives and barbiturates. We will also exclude current smokers because of the known effects of tobacco use on proinflammatory cytokine levels. (Helen, I would suggest to remove this sentence. It is clear from studies that patients are higher risk for susceptibility and increased disease activity with smoking. It may decrease our enrollment.)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-11; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lavretsky, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States

REFERENCES:
- See also: Milnacipran for Treatment of Pain in Older Adults With Rheumatoid Arthritis — http://www.semel.ucla.edu/latelife

RESULTS

PARTICIPANT FLOW:
Groups:
- Milnacipran, Active Drug, Open-label: All subjects will be free of antidepressant medications or opiates, or any other medications used to treat pain for at least 2 weeks prior to initiation of dose titration. Patients will be allowed to escalate up to 100 mg a day, or to their maximum tolerated dose in the course of the first week. The stable-dose phase will be a 10-week period during which patients will take medications at the final dose achieved (either 100 mg per day in divided doses, or the maximum tolerated dose of less than 100 mg per day). Final efficacy assessments will be made at the termination visit, and the study medication will be tapered down following 12 weeks of drug treatment.
  Milnacipran: All subjects will be free of antidepressant medications or opiates, or any other medications used to treat pain for at least 2 weeks prior to initiation of dose titration. Patients will be allowed to escalate up to 100 mg a day: Day 1: 12.5 mg once a day; Days 2-3: 25 mg/day (12.5 mg twice daily); Days 4-7: 50 mg/day
Period: Overall Study
Arm/Group | Milnacipran, Active Drug, Open-label
Started | 18
Completed | 12
Not Completed | 6
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Groups:
- Milnacipran, Active Drug, Open-label: All subjects will be free of antidepressant medications or opiates, or any other medications used to treat pain for at least 2 weeks prior to initiation of dose titration. Subjects will be allowed to escalate up to 100 mg a day or to their maximum tolerated dose in the course of the first week: Day 1: 12.5 mg once a day; Days 2-3: 25 mg/day (12.5 mg twice daily); Days 4-7: 50 mg/day (25 mg twice daily); After Day 7: 100 mg/day (50 mg twice daily). The stable-dose phase will be a 10-week period during which patients will take medications at the final dose achieved (either 100 mg per day in divided doses, or the maximum tolerated dose of less than 100 mg per day). Final efficacy assessments will be made at the termination visit, and the study medication will be tapered down following 12 weeks of drug treatment.
Arm/Group | Milnacipran, Active Drug, Open-label
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 67.5 [58 to 89]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Pain Rating Index
Description: The Pain Rating Index ranked values associated with adjectives depicting the severity of pain from the McGill Pain Questionnaire (MPQ). The assessment is comprised of 15 adjectives, each of which is scored on a scale ranging from 0 (none) to 3 (severe) and summed to arrive at a score ranging from 0 (no pain) to 45 (worst possible pain), to measure the extent of pain/tenderness and swelling. The Pain Rating Index final scores were averaged to indicate an overall report of joint pain and stiffness.
Time Frame: Change score at baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipran, Active Drug, Open-label
Number analyzed (Participants) | 12
units on a scale | -3.7 (6.6)

2. Secondary Outcome: Visual Analogue Scale to Evaluate Fatigue (VAS-F)
Description: The Visual Analogue Scale to Evaluate Fatigue (VAS-F) is an assessment of fatigue severity. The Visual Analogue Scale (VAS) measures a characteristic or attitude that ranges across a continuum of values from none (0) to an extreme amount of fatigue and energy (10). Scores fall between 0 and 10 anchored by word descriptors at each end and the patient marks on the line the point that they feel represents their perception of their current state. The scale consists of 18 items relating to the subjective experience of fatigue. Two subscales are summed separately and reported as follows: Items 1-5 and 11-18 represent fatigue from none (0) to extreme fatigue (10) and items 6-10 represent energy from none (0) to extreme energy (10). The outcome measures the change scores of energy and fatigue from Week 1 to Week 12. The VAS subscales for Fatigue Scale range: 0-130 and Energy Scale range: 0-50 with higher scores indicating greater energy and fatigue.
Time Frame: Change scores from Week 1 to Week 12 of energy and fatigue
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipran, Active Drug, Open-label
Number analyzed (Participants) | 12
units on a scale
  Fatigue Subscale | 15.2 (18.9)
  Energy Subscale | 3.7 (16.4)

3. Secondary Outcome: (UKU) Side Effects Rating Scale Profile
Description: The UKU assessment will rate the number of participants with emerging adverse events.
Time Frame: Weeks 1-4, 6, 8, 10, 12
Measure: Count of Participants; unit: Participants
Arm/Group | Milnacipran, Active Drug, Open-label
Number analyzed (Participants) | 12
Participants
  Concentration difficulties | 1
  Asthenia / Lassitude / Increased Fatiguability | 6
  Sleepiness / Sedation | 2
  Failing Memory | 1
  Depression | 2
  Reduced Duration of Sleep | 1
  Nausea / Vomiting | 3
  Micturition Disturbances | 2
  Increased Tendency to Sweating | 3
  Ejaculatory Dysfunction | 1
  Tension Headache | 2

4. Secondary Outcome: Profile of Mood States (POMS)
Description: Depressive symptoms: Repeated assessment of depressive symptoms severity will be made using the Profile of Mood States (POMS). The scale consisted of 65 adjectives rated on 5-point scale 0= not at all; 1=a little; 2=moderately; 3=quite a bit; 4=extremely. Five subscales were included in analysis: tension-anxiety (9 items, score range: 0-36), depression (15 items, range 0-60), friendliness (12 items, range 0-48), vigor-activity (8 items, range 0-32), and fatigue (7 items, range 0-28). Higher vigor-activity and friendliness scores reflect a good mood or emotion (high scores indicating better outcomes), and low scores in the other subscales (tension, depression, and fatigue) reflect a good mood or emotion (low scores indicating better outcomes).
Time Frame: Week 1 and 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipran, Active Drug, Open-label
Number analyzed (Participants) | 12
units on a scale
  POMS Anxiety Week 1 | 5.75 (5.12)
  POMS Depression Week 1 | 4.08 (3.60)
  POMS Vigor Week 1 | 13.00 (6.03)
  POMS Fatigue Week 1 | 6.67 (6.27)
  POMS Friendliness Week 1 | 6.42 (3.82)
  POMS Anxiety Week 12 | 5.50 (4.56)
  POMS Depression Week 12 | 3.92 (6.64)
  POMS Vigor Week 12 | 16.83 (5.92)
  POMS Fatigue Week 12 | 6.00 (4.86)
  POMS Friendliness Week 12 | 9.42 (5.99)

5. Secondary Outcome: Connor-Davidson Resilience Scale (CD-RISC)
Description: Resilience: the Connor-Davidson Resilience scale (CD-RISC) quantifies stress coping ability. The CD-RISC is a 25-item self-administered scale, although where necessary, a staff professional could read out each question to the subject and record the answer. The subject is directed to respond to each question with reference to the previous month, understanding that if a particular situation has not arisen in this time, then the response should be determined by how the person thinks they would have reacted. Scoring of the full 25 item scale is based on summing the total of each item, which is scored from 0-4. The full range is therefore from 0 to 100, with higher scores reflecting greater resilience. The outcome measure is a change score from Week 1 to Week 12.
Time Frame: Change Scores from Week 1 to Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipran, Active Drug, Open-label
Number analyzed (Participants) | 12
units on a scale | -2.2 (8.0)

ADVERSE EVENTS:
Arm/Group | Milnacipran, Active Drug, Open-label
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 6/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Milnacipran, Active Drug, Open-label (N=18)
Nausea (Gastrointestinal disorders) | 3
Concentration Difficulties (Psychiatric disorders) | 1
Asthenia (Psychiatric disorders) | 6
Sleepiness / Sedation (Psychiatric disorders) | 2
Failing Memory (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Reduced Duration of Sleep (Psychiatric disorders) | 1
Micturition Disturbances (Renal and urinary disorders) | 2
Increased Tendency to Sweat (Nervous system disorders) | 3
Ejaculatory Dysfunction (Reproductive system and breast disorders) | 1
Tension Headache (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No